CLINICAL TRIAL: NCT04471038
Title: A Phase 1, Randomized Double-Blind, Placebo-Controlled, Single Ascending Dose Safety, Tolerability, and Pharmacokinetics Study of SAB-176 in Healthy Adults
Brief Title: Safety, Tolerability, and Pharmacokinetics of SAB-176 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SAb Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAB-176-101
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Influenza Type A; Influenza Type B; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, placebo-controlled dose-escalating cohort design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 1 mg/mL SAB-176 in normal (0.9%) Saline; concentration 1 mg/mL (0.1%)
  Interventions: Biological: SAB-176
- Cohort 2 (Experimental): 10 mg/kgSAB-176 in normal (0.9%) Saline; concentration 4 mg/mL (0.4%)
  Interventions: Biological: SAB-176
- Cohort 3 (Experimental): 25 mg/kgSAB-176 in normal (0.9%) Saline; concentration 20 mg/mL (2.0%)
  Interventions: Biological: SAB-176
- Cohort 4 (Experimental): 50 mg/kg SAB-176 in normal (0.9%) Saline; concentration 20 mg/mL (2.0%)
  Interventions: Biological: SAB-176
- Cohort 5 (Placebo Comparator): Normal (0.9%) saline in approximately the same volume as each cohort in the experimental drug arm.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: SAB-176 — Anti-Influenza Human Immunoglobulin Intravenous (Tc bovine derived)
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4
Other: Normal Saline — Normal (0.9%) saline in approximately the same volume as each cohort in the experimental drug arm
  Arms: Cohort 5

SUMMARY:
Influenza causes substantial morbidity and mortality worldwide despite available antivirals and vaccines. SAB Biotherapeutics, Inc. has developed SAB-176, an anti-influenza human immunoglobulin (transchromosomic [Tc] bovine-derived) intravenous therapeutic to treat past and current strains of Type A Influenza and Type B Influenza. This study will evaluate the safety, tolerability, and pharmacokinetics of SAB-176 in healthy participants.

DETAILED DESCRIPTION:
This safety and tolerability study of IV SAB-176 consisted of up to 4 single dose levels or cohorts (Cohort 1 through 4) in a double-blind, randomized, placebo-controlled dose-escalating cohort design. Four cohorts of 3 to10 subjects each were administered a single IV dose of SAB-176 or saline placebo. At very low doses, the concern was primarily allergic or T-cell activation/cytokine storm, so small cohort sizes were utilized. As the target dose was approached, the sample size was increased to increase the likelihood of detecting toxicity events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤60 years
2. Body mass index (BMI) of 19-32 kg/m2
3. Subjects must have values in normal ranges for basic labs (i.e., CBC, PT/INR, Chem-7, and LFTs), unless deemed not clinically significant by the PI.
4. Estimated glomerular filtration rate ≥90 mL/min at screening, calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
5. Subjects must agree to:

Not take any prescription or over-the-counter (OTC) medications with the exception of acetaminophen, ibuprofen, vitamins, seasonal allergy medications, and/or contraceptive medications, or others unless approved by the study investigator, for a period 7 days prior to study drug administration (i.e., Day 0). Use one of the following in order to avoid pregnancy: Females who are able to become pregnant (i.e., are not postmenopausal, have not undergone surgical sterilization, and are sexually active with men) must agree to use at least 2 effective forms of contraception from the date of the subject's signing of the informed consent form through 60 days after the last dose of study drug. At least one of the methods of contraception should be a barrier method.

Males who have not undergone surgical sterilization and are sexually active with women must agree to use condoms plus have a partner use at least one additional effective form of contraception from the date of the subject's signing of the informed consent form through 60 days after the last dose of study drug.

Neither females or males should donate oocysts or sperm for use in artificial insemination through 60 days after the last dose of study drug.

Exclusion Criteria:

1. Any history of allergy, anaphylaxis, or severe reaction to beef products (including milk and gelatin)
2. Any history of allergy, anaphylaxis, or severe reaction to IVIg or human blood products
3. Any chronic medical problem/condition that require medications needed to maintain the subject's health. Exceptions to this restriction can be allowed for minor health conditions that are treated with Tylenol, over-the-counter non-steroidal anti-inflammatories, vitamins, seasonal allergy medications, or oral/transdermal/IUD contraceptives, etc. The study investigator will make a determination to exclude a subject based upon their medical history and the type and frequency of the drug substance.
4. History of cardiovascular disease, cardiomyopathy, heart failure, or unexplained syncope
5. Abnormal clinically significant 12-lead electrocardiogram (ECG), per PI discretion
6. Subjects who have been laboratory confirmed or clinically diagnosed with influenza within seven days prior to infusion (by subject history) will be deferred from infusion. Any subject with signs and symptoms of an active respiratory infection on the day of infusion will be deferred until the infection is cleared in the opinion of the investigator. Subjects that present with an active upper respiratory infection on the day of infusion will be tested with an FDA licensed Influenza A/B Antigen Test. Signs and symptoms constituting an upper respiratory infection include cough, sore throat, or rhinorrhea with or without fever.
7. Enrollment will be delayed for all patients who have other intercurrent infections (e.g., gastroenteritis, abscess, etc.).
8. Women who are breast-feeding
9. Positive urine or serum pregnancy test
10. Positive urine drug screen (UDS)
11. Clinically significant results, including laboratory results, as determined by study investigator
12. Positive rheumatoid factor
13. IgA deficiency (defined as IgA less than 7 mg/dL)
14. Participation in another research study with receipt of any investigational drug within 5 half-lives or 30 days, whichever is longer, prior to study drug administration (i.e., Day 0) and until completion of the study
15. Participation in any other research study until the completion of the study
16. Receipt of blood products within 2 months prior to study drug administration (i.e.Day 0)
17. Receipt of any vaccination within 30 days prior to study drug administration (i.e.Day 0)
18. Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca N Wood-Horrall, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD, Phase 1 Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification (test, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication and ending 36 months following article publication
Access Criteria: Anyone who wishes to access the data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 2 | 4 | 6 | 8 | 7
Completed | 2 | 4 | 6 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 2 | 4 | 6 | 8 | 7 | 27
Age, Customized [Mean (Standard Deviation); unit: years] | 29.0 (5.66) | 43.3 (14.41) | 40.5 (10.07) | 34.1 (7.72) | 35.7 (9.95) | 36.9 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 2 | 4 | 13
  Male | 0 | 1 | 4 | 6 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 4 | 4 | 15
  Not Hispanic or Latino | 0 | 2 | 3 | 4 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 1 | 0 | 5
  White | 1 | 2 | 4 | 7 | 7 | 21
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Screening Weight (kg) [Mean (Standard Deviation); unit: kg] | 76.10 (18.950) | 62.68 (11.054) | 85.95 (18.888) | 85.26 (10.859) | 72.67 (11.226) | 78.13 (15.242)
Screening BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.70 (0.707) | 23.95 (4.779) | 27.95 (3.500) | 28.58 (2.230) | 26.13 (4.389) | 27.13 (3.689)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Having Adverse Events
Description: Incidence and severity of other adverse events and severe adverse events (SAE)
Time Frame: 90 days
Population: At each level of subject summarization, a subject is counted once if the subject reported one or more events.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 4 | 6 | 8 | 7
Participants | 0 | 1 | 1 | 1 | 2

2. Secondary Outcome: Number of Participants With Anti-SAB-176 Antibodies Elicited by SAB-176
Description: Number of subjects showing antidrug antibodies to SAB-176 through day 90
Time Frame: 90 Days
Population: Subjects who received SAB-176 or placebo with 1 or more samples obtained after SAB-176 or placebo administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 2 | 4 | 6 | 8 | 0
Participants | 0 | 0 | 2 | 1 |

ADVERSE EVENTS:
Time Frame: AEs that occur following enrollment of the subject (by signing the informed consent) through the follow up period at Day 90.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/6 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/6 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/2 | 1/4 | 1/6 | 1/8 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=2) | Cohort 2 (N=4) | Cohort 3 (N=6) | Cohort 4 (N=8) | Cohort 5 (N=7)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthemia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular skeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT04471038/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT04471038/SAP_001.pdf